CLINICAL TRIAL: NCT04299815
Title: Lactate in the Gut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1-10-72-8-20
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-02

CONDITIONS: Lactate; Healthy; Hyperlactatemia
Keywords: lactate; metabolism; Gastric emptying; GDF-15; insulin; incretin hormones
MeSH Terms: conditions — Hyperlactatemia; Insulin Resistance | interventions — Sodium Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral lactate (Active Comparator): Sodium D/L lactate solution, 25g/L in 300mL water
  Interventions: Drug: Oral Sodium Lactate
- Iso-lactic intravenous lactate infusion (Placebo Comparator): iv sodium D/L lactate to elevate [lactate] to the same levels as measured on day 1 + oral sodium chloride, 300 mL
  Interventions: Drug: Intravenous sodium lactate

INTERVENTIONS:
Drug: Oral Sodium Lactate — 25 grams of D/L lactate dissolved in 300mL water.
  Arms: Oral lactate
Drug: Intravenous sodium lactate — intravenous sodium lactate + oral sodium-chlorid solution
  Arms: Iso-lactic intravenous lactate infusion

SUMMARY:
Lactate is formed naturally in the body in example during physical activity. However, lactate is also formed during food fermentation where certain bacterial strains form lactate. Lactate can also be produced chemically. An example of this is Ringer-lactate which is used for volume replacement when treating dehydrated patients.

As a source of carbon-molecules, lactate is believed to be an important oxidative fuel source in all major organs and yields adenosine triphosphate (ATP) production through Krebs cycle, the Electron Transport Chain in the mitochondria as well as by being a key precursor for gluconeogenesis.

Metformin is the first drug of choice for type 2 diabetes treatment. Use of metformin often results in a small but significant weight loss in overweight users. It is known that metformin increases the lactate concentration in the gut. It is also known also know that metformin use is associated with an increase in blood concentrations of growth differentiation factor 15 (GDF-15). Receptors for GDF-15 can be found in parts of the brain associated with control of appetite. In rats increases in [GDF-15] results in a decrease in appetite and thus weight loss. GDF-15 is thought to be involved in the normal energy homeostasis.

With this study the investigators want to examine the hormonal, metabolic and mechanical effects of lactate in the gut in healthy volunteers. Our hypothesis is that lactate has beneficial effects which may be though an increase in GDF-15 in the blood.

Volunteers will undergo two study days separated by at least 7 days and a maximum of 1 month.

* On day one volunteers will drink a sodium-lactate solution (intervention). The investigators will also administrate 1500mg paracetamol to assess gastric emptying and do blood samples over 4 hours. The investigators measure [lactate] every 15 min. Every hour the investigators will ask volunteers questions regarding hunger and thoughts of future food intake (questionnaire). After 4 hours of blood sampling the investigators will serve volunteers an all-you-can-eat meal of sandwich and measure how must they ate.
* On day two volunteers will drink a sodium chloride solution. Furthermore, the investigators administrate intravenous D/L sodium lactate in order to reach the same plasma [lactate] on day 2 as was done on day 1. The rest of day two is identical to day 1.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Age 18-50 years
* BMI 20-30 kg/m2
* In good health with no daily use of prescription medicine based on medical history, clinical examination and blood samples.
* Spoken and written informed consent

Exclusion Criteria:

* Chronic illness or daily use of prescription medicine .
* Abnormal screening blood samples as judged by the PI
* Does not understand or speak Danish

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
GDF-15 | 4 hours
  Difference in [GDF-15] between intervention and placebo

SECONDARY OUTCOMES:
glucagon-like peptide -1 | 4 hours
  Difference in [glucagon-like peptide -1] between intervention and placebo
Gastric inhibitory peptide (GIP) | 4 hours
  Difference in plasma [GIP] between intervention and placebo
free fatty acid | 4 hours
  Difference in [free fatty acid ] between intervention and placebo
cholecystokinin | 4 hours
  Difference in [cholecystokinin] between intervention and placebo
Ghrelin | 4 hours
  Difference in [Ghrelin] between intervention and placebo
Gastrin | 4 hours
  Difference in [Gastrin] between intervention and placebo
C-peptide | 4 hours
  Difference in [C-peptide] between intervention and placebo
glucose | 4 hours
  Difference in [glucose] between intervention and placebo
gastric emptying | 4 hours
  [Paracetamol] to asses gastric emptying
Evaluation of hunger | 4 hours
  Evaluation of hunger, thoughts of future food intake ect using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaj Rittig, postdoc, Study Chair — Steno Diabetes Center Aarhus (SDCA), Aarhus universitetshospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Pedersen MGB, Lauritzen ES, Svart MV, Stoy J, Sondergaard E, Thomsen HH, Kampmann U, Bjerre M, Jessen N, Moller N, Rittig N. Nutrient sensing: LEAP2 concentration in response to fasting, glucose, lactate, and beta-hydroxybutyrate in healthy young males. Am J Clin Nutr. 2023 Dec;118(6):1091-1098. doi: 10.1016/j.ajcnut.2023.10.007. Epub 2023 Oct 14. PMID 37844838
- [Derived] Pedersen MGB, Sondergaard E, Nielsen CB, Johannsen M, Gormsen LC, Moller N, Jessen N, Rittig N. Oral lactate slows gastric emptying and suppresses appetite in young males. Clin Nutr. 2022 Feb;41(2):517-525. doi: 10.1016/j.clnu.2021.12.032. Epub 2021 Dec 24. PMID 35016146